CLINICAL TRIAL: NCT01944020
Title: Effects of CPAP on Diet, Physical Activity, and Cardiovascular Risk
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Ari Shechter, Assistant Professor of Medical Sciences, Columbia University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AAAO2006; 15SDG22680012 (Other Grant/Funding Number: American Heart Association)
Record Dates: First submitted 2013-09-12; First posted 2013-09-17 (Estimated); Results first posted 2022-05-03 (Actual); Last update posted 2022-05-03 (Actual); Status verified 2022-04

CONDITIONS: Sleep Apnea Syndromes
Keywords: Sleep Apnea, Obstructive; Energy Balance; Food Intake; Energy Expenditure; Sleep; Obesity
MeSH Terms: conditions — Sleep Apnea Syndromes; Sleep Apnea, Obstructive; Obesity

STUDY DESIGN:
Intervention Model Description: treatment group: individuals with OSA using CPAP control group: individuals with OSA not using CPAP
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention - CPAP use (Experimental): Active CPAP will be a therapeutic dose of positive airway pressure each night for 2 months
  Interventions: Device: CPAP
- Control - No CPAP use (No Intervention): Control will be no use of CPAP for 2 months

INTERVENTIONS:
Device: CPAP — use of CPAP each night for 2 months
  Arms: Intervention - CPAP use

SUMMARY:
Obstructive sleep apnea (OSA) is characterized by recurrent episodes of partial or complete loss of airflow during sleep, due to narrowing or closure of the upper airway. The resulting hypoxia has many cardiometabolic consequences, and leads to a disruption of sleep quality including reductions in the expression of rapid eye movement (REM) sleep and slow wave sleep (SWS). Patients also frequently experience excessive daytime sleepiness (EDS), which, when present with OSA, defines the clinical entity OSA syndrome (OSAS). Obesity is the leading risk factor for the development of OSA. Interestingly, it has been suggested that the disorder itself may contribute to further weight gain, presenting a vicious cycle wherein OSA and obesity perpetuate each other. OSAS may promote weight gain by placing patients in a state of positive energy balance characterized by low levels of physical activity and disrupted patterns of appetite-regulating hormones. Continuous positive airway pressure (CPAP), the gold-standard treatment of OSAS, may improve energy balance in these patients, although this has not yet been adequately studied. The current proposal will investigate the effects of 2 months of CPAP on energy balance and cardiovascular risk in obese patients with OSA. Patients will be instructed to use CPAP at home each night throughout the 2-month treatment phases. At baseline and at the conclusion of the 2-month treatment phase, the investigators will measure levels of free-living physical activity, sleepiness, sleep quality, body composition, cardiovascular risk factors, appetite-regulating hormones, hunger, and ad libitum food intake. There will also be a control group with OSA individuals studied at baseline and again after 2 months with no CPAP use. It is hypothesized that CPAP compared to no treatment treatment will result in improvements in energy balance, including increased physical activity, reductions in abnormally high levels of circulating leptin levels, and reductions in hunger, food intake, and cardiovascular risk factors. These improvements are hypothesized to be associated with increases in the expression of REM sleep and SWS, and reduced EDS as a result of CPAP.

DETAILED DESCRIPTION:
This study investigates the effects of 2 mo of continuous positive airway pressure (CPAP) on physical activity, energy intake (EI), and cardiovascular risk factors in overweight/obese patients with obstructive sleep apnea (OSA).

Patients will be instructed to use CPAP at home each night throughout the 2 mo treatment phase. Before and after the 2 mo treatment phase, patients will undergo a 1-d in-lab testing period at the Clinical Research Resource (CRR) at Columbia University Medical Center. Upon completion of the laboratory phase 1, patients will return home for a 2 mo treatment period, followed by the second tracking period including laboratory visit 2.

Before and at the conclusion of the 2 mo treatment phase, patients will enter the laboratory at the Columbia University Medical Center for a 1-d period. Patients will arrive at ~0800 h and will remain in the laboratory for the following 24 h. Blood will be sampled in the fasting state in the morning, and will be assayed for select appetite-regulating hormones (leptin, ghrelin, adiponectin, glucagon-like peptide-1). We will also assess body composition. During the laboratory day, ad libitum EI will be measured for each treatment phase. Breakfast, lunch, snack, and dinner will be served at the standard times, but each meal item will be served in excess such that patients will be able to eat as much or as little of each food as they choose. Additional snack choices will also be freely available during the wake episode.

There will also be a control group of individuals with OSA who do not use CPAP who are studied at baseline and again after a 2 month period in procedures similar to those undergoing treatment.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of obstructive sleep apnea (OSA) and excessive daytime sleepiness (EDS)
* body mass index of at least 25 kg/m^2

Exclusion Criteria:

* prior treatment with CPAP
* shift workers
* type 2 diabetes
* poorly controlled severe hypertension
* anemia
* history of coronary artery disease, transient ischemic attack, stroke
* currently taking anti-psychotic, anti-depressive, or hypnotic medications
* females currently taking hormone replacement therapy
* females who are pregnant or have given birth within 1 year

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2015-05; Primary Completion 2018-09 (Actual); Study Completion 2018-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ari Shechter, Ph.D., Principal Investigator — New York Obesity Research Center, Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

REFERENCES:
- [Derived] Shechter A, Kovtun K, St-Onge MP. Effects of continuous positive airway pressure on energy intake in obstructive sleep apnea: A pilot sham-controlled study. Physiol Behav. 2016 Dec 1;167:399-403. doi: 10.1016/j.physbeh.2016.10.011. Epub 2016 Oct 18. PMID 27769851
- [Derived] Shechter A, Pham T, Rising R, St-Onge MP. Effects of CPAP on energy expenditure in obese obstructive sleep apnoea patients: A pilot study. Obes Res Clin Pract. 2015 Nov-Dec;9(6):618-21. doi: 10.1016/j.orcp.2015.08.015. Epub 2015 Sep 11. PMID 26371702

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention - CPAP Use | Control - No CPAP Use
Started | 17 | 12
Completed | 12 | 12
Not Completed | 5 | 0
Not completed — Withdrawal by Subject | 5 | 0

BASELINE CHARACTERISTICS:
Population: Participants who completed the intervention
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention - CPAP Use | Control - No CPAP Use | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.7 (10.9) | 53.1 (11.6) | 50.4 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 10
  Male | 7 | 7 | 14
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White Non-Hispanic | 5 | 0 | 5
  Black Non-Hispanic | 4 | 8 | 12
  Asian Non-Hispanic | 1 | 1 | 2
  Hispanic | 2 | 3 | 5
Region of Enrollment [Number; unit: participants]
  United States | 12 | 12 | 24
Body mass index [Mean (Standard Deviation); unit: kg/m^2] | 35.6 (4) | 34.9 (6.5) | 35.2 (5.2)

OUTCOME MEASURES:

1. Primary Outcome: Fat Mass (% of Total Body Mass)
Description: Fat mass (% of total body mass) measured via BODPOD at baseline preceding treatment phase, and at the end of treatment phase.
Time Frame: At baseline ("Pre") and after 2 months of treatment ("Post") or control
Population: all completed CPAP group and non-CPAP group participants
Measure: Mean (Standard Deviation); unit: percentage of total body mass
Arm/Group | Intervention - CPAP Use | Control - No CPAP Use
Number analyzed (Participants) | 12 | 12
percentage of total body mass
  Pre (i.e., at baseline) | 40.0 (7.6) | 37.7 (11.2)
  Post (i.e., after 2 months of treatment) | 38.7 (7.3) | 38.6 (10.4)

2. Secondary Outcome: ad Libitum Food Intake (Total Daily Calories Consumed)
Description: Participants will be served meals (breakfast, lunch, dinner, snack) at specified times, but food will be served in excess such that participants will be able to eat as much as they want.
Time Frame: At baseline ("Pre") and after 2 months ("Post") of treatment or control
Population: Data from 1 participant in the Active CPAP group were missing from analyses due to technical problem.
Measure: Mean (Standard Deviation); unit: kcal
Arm/Group | Intervention - CPAP Use | Control - No CPAP Use
Number analyzed (Participants) | 11 | 12
kcal
  Pre (at baseline) | 2999.9 (967.8) | 4631.0 (1854.5)
  Post (after 2 months) | 3301.6 (773.1) | 4479.3 (1769.4)

3. Other Pre Specified Outcome: Appetite-regulating Hormones and Cardiovascular Risk Factors at 2 Months
Description: Blood will be sampled once in the morning in the fasted state to assay levels of circulating hormones that regulate appetite and hunger, including leptin, ghrelin, adiponectin, and glucagon-like peptide-1, as well as inflammatory and cardiovascular risk markers
Time Frame: At baseline and after 2 months of treatment or control
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 2 months
Description: any side effect of adverse event
Arm/Group | Intervention - CPAP Use | Control - No CPAP Use
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 0/12 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-09-29): https://cdn.clinicaltrials.gov/large-docs/20/NCT01944020/Prot_SAP_000.pdf
  • Informed Consent Form (2021-07-03): https://cdn.clinicaltrials.gov/large-docs/20/NCT01944020/ICF_001.pdf